CLINICAL TRIAL: NCT00607087
Title: Effect of Insulin Glulisine Compared to Insulin Aspart and Insulin Lispro When Administered by Continuous Subcutaneous Insulin Infusion (CSII) on Specific Pump Parameters in Patient With Type 1 Diabetes Mellitus
Acronym: PUMP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: APIDR_C_02083; 2007-003579-38 (EudraCT Number)
Record Dates: First submitted 2008-01-23; First posted 2008-02-05 (Estimated); Results first posted 2010-07-30 (Estimated); Last update posted 2010-08-31 (Estimated); Status verified 2010-08

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — insulin glulisine; Insulin Lispro; Insulin Aspart

ARMS (3):
- sequence 1 (Experimental): sequence 1: insulin glulisine / insulin aspart / insulin lispro.
  Interventions: Drug: Insulin glulisine; Drug: Insulin lispro; Drug: Insulin aspart
- Sequence 2 (Experimental): Sequence 2: insulin aspart / insulin lispro / insulin glulisine
  Interventions: Drug: Insulin glulisine; Drug: Insulin lispro; Drug: Insulin aspart
- Sequence 3 (Experimental): Sequence 3: insulin lispro / insulin glulisine / insulin aspart
  Interventions: Drug: Insulin glulisine; Drug: Insulin lispro; Drug: Insulin aspart

INTERVENTIONS:
Drug: Insulin glulisine — 100 U/ml, administration by Continuous Subcutaneous Insulin Infusion with external pump
Drug: Insulin lispro — 100 U/ml, administration by Continuous Subcutaneous Insulin Infusion with external pump
Drug: Insulin aspart — 100 U/ml, administration by Continuous Subcutaneous Insulin Infusion with external pump

SUMMARY:
Primary objective: To demonstrate the superiority of insulin glulisine over insulin aspart and insulin lispro administered by external pump in term of unexplained hyperglycemia and/or infusion set occlusion.

Main Secondary objectives:

To compare insulin glulisine, insulin aspart and insulin lispro on:

* Unexplained hyperglycemia
* Infusion set occlusion
* Hypoglycemic episodes,7-point blood glucose profiles
* Episodes of significant ketosis and/or risk level for impending diabetic ketoacidosis
* Time to change the infusion set
* HbA1c (Glycosylated hemoglobin)
* Overall safety: incidence of adverse events

DETAILED DESCRIPTION:
The maximal duration of the study participation for patients was 41 weeks and one day, split in:

* a 2-week screening period,
* a 39-week treatment period: 3 treatment periods of 13 weeks with a crossover alternative regimen, including a dose adjustment period of 1 week at the beginning of each period (sequence1: insulin glulisine, then insulin aspart, then insulin lispro; sequence2: insulin aspart, then insulin lispro, then insulin glulisine; sequence 3: insulin lispro, then insulin glulisine, then insulin aspart)
* and a follow-up period of 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetic subjects
* Treated with insulin for at least 2 years and by CSII for at least 6 months
* Using the same insulin (insulin glulisine, insulin aspart or insulin lispro) in CSII for at least 3 months with the same external pump compatible with the 3 short acting insulin analogues used in the study
* Using the same type of infusion set (catheter and cannula) for at least 3 months
* Performing at least 3 blood glucose controls per day
* HbA1c < 8.5%
* Body mass index (BMI) < 35 kg/m²
* Ability and willingness to perform blood glucose and ketone monitoring using the Sponsor-provided combined glucose and ketone meter and patient diary at home

Exclusion Criteria:

* Diabetes other than Type 1
* Total daily dose of insulin greater than 90 U/day
* Using an insulin pump requiring pre-filled cartridges
* History of infection at infusion site requiring a drainage in the last 3 months
* History of severe episodes of ketosis requiring hospitalization in the last 6 months
* Active proliferative retinopathy, as defined by a photocoagulation or vitrectomy occurrence in the 6 months prior to visit 1, or any other unstable (rapidly progressing) retinopathy that may require photocoagulation or surgical treatment during the study. An ophthalmoscopic examination should have been performed in the 2 years prior to study entry
* Pregnancy (women of childbearing potential must have a negative pregnancy test at study entry and a medically approved contraception method) or breastfeeding
* Treatment with systemic corticosteroids or medication known to influence insulin sensitivity in the 3 months prior to visit 1
* Treatment with antidiabetic drug other than insulin in the 3 months prior to visit 1
* Likelihood of requiring treatments during the study which are not permitted
* Treatment with an investigational product in the 30 days prior to visit 1
* History of sensitivity to the study drugs or to drugs with a similar chemical structure
* Presence of any condition (medical, including clinically significant abnormal laboratory test, psychological, social or geographical) actual or anticipated that the Investigator feels would compromise the patient safety or limit his/her successful participation in the study
* Night shift workers
* Impaired renal function as shown by serum creatinine ≥1.5 mg/dL (133 μmol/L) or ≥1.4 mg/dL (124 μmol/L) in men and women, respectively
* Impaired hepatic function as shown by Alanine aminotransferase (ALT) and/or Aspart aminotransferase (AST) greater than three times the upper limit of normal range)
* Alcohol or drug abuse in the last year
* Mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2008-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs, Study Director — Sanofi
Locations (12):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Macquarie Park, Australia
- Sanofi-Aventis Administrative Office, Vienna, Austria
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Netanya, Israel
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, PE Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Seoul, South Korea
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Bromma, Sweden
- Sanofi-Aventis Administrative Office, Guildford Surrey, United Kingdom

REFERENCES:
- [Derived] van Bon AC, Bode BW, Sert-Langeron C, DeVries JH, Charpentier G. Insulin glulisine compared to insulin aspart and to insulin lispro administered by continuous subcutaneous insulin infusion in patients with type 1 diabetes: a randomized controlled trial. Diabetes Technol Ther. 2011 Jun;13(6):607-14. doi: 10.1089/dia.2010.0224. Epub 2011 Apr 2. PMID 21457066

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Multicenter study: 44 active centers from 12 countries in Europe, USA and Asia Pacific region. Study Initiation date: January 8, 2008, Study Completion Date: June 15, 2009.
Pre-assignment Details: 359 participants screened; 289 randomized; 288 patients treated (1 patient not treated per physician's decision): 274 with insulin glulisine, 269 with insulin lispro, 266 with insulin aspart.
  The safety population, (N=288 patients randomized and treated) is described in the participant flow and baseline characteristics.
Groups:
- Sequence 1: insulin glulisine / insulin aspart / insulin lispro
- Sequence 2: insulin aspart / insulin lispro / insulin glulisine
- Sequence 3: insulin lispro / insulin glulisine / insulin aspart
Period: Overall Study
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3
Started | 99 | 95 | 94
Completed | 84 | 84 | 84
Not Completed | 15 | 11 | 10
Not completed — Withdrawal by Subject | 9 | 4 | 4
Not completed — Adverse Event | 3 | 2 | 3
Not completed — Other reason | 1 | 5 | 2
Not completed — Poor compliance to protocol | 1 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0
Period: Period 1
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3
Started | 99 | 95 | 94
Completed | 87 | 89 | 89
Not Completed | 12 | 6 | 5
Not completed — Withdrawal by Subject | 7 | 2 | 3
Not completed — Adverse Event | 3 | 0 | 0
Not completed — Poor compliance to protocol | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Other reason | 0 | 4 | 2
Period: Period 2
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3
Started | 87 | 89 | 89
Completed | 86 | 86 | 84
Not Completed | 1 | 3 | 5
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Other reason | 1 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 3
Not completed — Poor compliance to protocol | 0 | 0 | 1
Period: Period 3
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3
Started | 86 | 86 | 84
Completed | 84 | 84 | 84
Not Completed | 2 | 2 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 99 | 95 | 94 | 288
Age Continuous [Mean (Standard Deviation); unit: years] | 43.45 (13.71) | 45.84 (13.59) | 44.04 (12.87) | 44.43 (13.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 54 | 48 | 151
  Male | 50 | 41 | 46 | 137
Region of Enrollment [Number; unit: participants]
  United States | 22 | 21 | 21 | 64
  France | 8 | 9 | 10 | 27
  Hungary | 4 | 4 | 6 | 14
  Spain | 11 | 9 | 10 | 30
  Austria | 7 | 9 | 8 | 24
  Australia | 4 | 4 | 3 | 11
  Israel | 11 | 11 | 10 | 32
  Netherlands | 8 | 8 | 7 | 23
  United Kingdom | 5 | 4 | 4 | 13
  Italy | 9 | 7 | 7 | 23
  Sweden | 9 | 8 | 7 | 24
  Korea, Republic of | 1 | 1 | 1 | 3
Previous insulin at study entry [Number; unit: participants] — Total patients analyzed n=287 due to one missing data in the "sequence 2" group
  participants
    Insulin glulisine | 4 | 2 | 2 | 8
    Insulin aspart | 32 | 43 | 42 | 117
    Insulin lispro | 63 | 49 | 50 | 162
Duration of treatment with previous insulin at study entry [Mean (Standard Deviation); unit: years] — Total patients analyzed n=286 due to one missing data in the "sequence 1" and in the "sequence 2" groups
  years | 4.84 (3.58) | 4.37 (3.05) | 4.79 (3.00) | 4.67 (3.22)
Duration of treatment with insulin at study entry [Mean (Standard Deviation); unit: years] | 22.39 (13.53) | 23.07 (13.33) | 22.75 (11.08) | 22.73 (12.67)
Total daily bolus insulin dose [Mean (Standard Deviation); unit: Units] — Total patients analyzed n=285 due to 3 missing data: 2 in the "sequence 1" and 1 in the "sequence 2" groups
  Units | 19.61 (9.40) | 18.58 (10.34) | 19.35 (7.78) | 19.18 (9.22)
Duration of treatment with CSII (continuous subcutaneous insulin infusion) at study entry [Mean (Standard Deviation); unit: years] | 5.99 (4.83) | 5.52 (5.27) | 6.31 (4.95) | 5.94 (5.01)
Total daily basal insulin infusion [Mean (Standard Deviation); unit: Units] — Total patients analyzed n=285 due to 3 missing data: 2 in the "sequence 1" and 1 in the "sequence 2" groups
  Units | 20.98 (8.84) | 19.99 (9.38) | 22.03 (9.17) | 21.00 (9.13)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] | 25.01 (3.53) | 25.25 (3.91) | 25.92 (3.98) | 25.39 (3.81)
Central fasting plasma glucose [Mean (Standard Deviation); unit: mg/dL] — Total patients analyzed n=284 due to 4 missing data: 2 in the "sequence 1" and 2 in the "sequence 3" groups
  mg/dL | 149.84 (59.03) | 147.45 (61.63) | 151.18 (64.06) | 149.48 (61.37)
Glycosylated Haemoglobin (HbA1c) [Mean (Standard Deviation); unit: Percent] | 7.38 (0.69) | 7.36 (0.61) | 7.41 (0.69) | 7.38 (0.66)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With at Least One Unexplained Hyperglycemia and/ or Confirmed Infusion Set Occlusion
Description: Unexplained hyperglycemia defined as blood glucose value above 300 mg/dL (16.7 mmol/L) with no apparent medical dietary, insulin dosage or pump failure reason.
  Pump infusion set occlusion defined by at least one of the following items:
  * pump occlusion alarm,
  * patient observation of an occlusion, spontaneously or because of elevated blood glucose value.
Time Frame: over 13 weeks of each treatment period
Population: Analysis was performed on the Intention To Treat (ITT) population. The Intent-To-Treat population is composed of all randomized patients having received the 3 insulins (Insulin glulisine, aspart and lispro) N=256 patients: (sequence 1: N=86, sequence 2: N=86; sequence 3: N=84 patients).
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Insulin Glulisine | Insulin Aspart | Insulin Lispro
Number analyzed (Participants) | 256 | 256 | 256
percentage of patients | 68.4 [62.7 to 74.1] | 62.1 [56.2 to 68.1] | 61.3 [55.4 to 67.3]
Statistical Analysis 1: Comparison: Insulin Glulisine vs Insulin Aspart; Test type: Superiority or Other; p = 0.039, McNemar — The p-value is adjusted for multiple comparisons. Each comparison is performed at the alpha level=2.5% (instead of 5%). Consequently a difference between 2 treatments is statistically significant if the corresponding p-value is <0.025
Statistical Analysis 2: Comparison: Insulin Glulisine vs Insulin Lispro; Test type: Superiority or Other; p = 0.031, McNemar — [p-value comment as in outcome 1, analysis 1]

2. Secondary Outcome: Monthly Rate of Unexplained Hyperglycemia and/ or Confirmed Infusion Set Occlusion
Description: as for outcome 1
Time Frame: over 13 weeks of each treatment period
Population: as for outcome 1
Measure: Mean (Standard Error); unit: events per patient per month
Arm/Group | Insulin Glulisine | Insulin Aspart | Insulin Lispro
Number analyzed (Participants) | 256 | 256 | 256
events per patient per month | 2.02 (0.15) | 1.32 (0.15) | 1.54 (0.15)
Statistical Analysis 1: Comparison: Insulin Glulisine vs Insulin Aspart; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Insulin Glulisine vs Insulin Lispro; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Patients With at Least One Unexplained Hyperglycemia
Description: Unexplained hyperglycemia defined as blood glucose value above 300 mg/dL (16.7 mmol/L) with no apparent medical dietary, insulin dosage or pump failure reason.
Time Frame: over 13 weeks of each treatment period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Insulin Glulisine | Insulin Aspart | Insulin Lispro
Number analyzed (Participants) | 256 | 256 | 256
percentage of patients | 61.3 [55.4 to 67.3] | 55.9 [49.8 to 61.9] | 56.3 [50.2 to 62.3]
Statistical Analysis 1: Comparison: Insulin Glulisine vs Insulin Aspart; Test type: Superiority or Other; p = 0.080, McNemar — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Insulin Glulisine vs Insulin Lispro; Test type: Superiority or Other; p = 0.107, McNemar — [p-value comment as in outcome 1, analysis 1]

4. Secondary Outcome: Monthly Rate of Unexplained Hyperglycemia
Time Frame: over 13 weeks of each treatment period
Population: as for outcome 1
Measure: Mean (Standard Error); unit: events per patient per month
Arm/Group | Insulin Glulisine | Insulin Aspart | Insulin Lispro
Number analyzed (Participants) | 256 | 256 | 256
events per patient per month | 1.61 (0.13) | 1.04 (0.13) | 1.23 (0.13)
Statistical Analysis 1: Comparison: Insulin Glulisine vs Insulin Aspart; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Insulin Glulisine vs Insulin Lispro; Test type: Superiority or Other; p < 0.001, McNemar — [p-value comment as in outcome 1, analysis 1]

5. Secondary Outcome: Percentage of Patients With at Least One Confirmed Infusion Set Occlusion
Description: Pump infusion set occlusion defined by at least one of the following items:
  * pump occlusion alarm,
  * patient observation of an occlusion, spontaneously or because of elevated blood glucose value.
Time Frame: over 13 weeks of each treatment period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Insulin Glulisine | Insulin Aspart | Insulin Lispro
Number analyzed (Participants) | 256 | 256 | 256
percentage of patients | 32.8 [27.1 to 38.6] | 27.0 [21.5 to 32.4] | 27.0 [21.5 to 32.4]
Statistical Analysis 1: Comparison: Insulin Glulisine vs Insulin Aspart; Test type: Superiority or Other; p = 0.079, McNemar — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Insulin Glulisine vs Insulin Lispro; Test type: Superiority or Other; p = 0.063, McNemar — [p-value comment as in outcome 1, analysis 1]

6. Secondary Outcome: Monthly Rate of Confirmed Infusion Set Occlusion
Time Frame: over 13 weeks of each treatment period
Population: as for outcome 1
Measure: Mean (Standard Error); unit: events per patient per month
Arm/Group | Insulin Glulisine | Insulin Aspart | Insulin Lispro
Number analyzed (Participants) | 256 | 256 | 256
events per patient per month | 0.41 (0.06) | 0.28 (0.06) | 0.31 (0.06)
Statistical Analysis 1: Comparison: Insulin Glulisine vs Insulin Aspart; Test type: Superiority or Other; p = 0.015, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Insulin Glulisine vs Insulin Lispro; Test type: Superiority or Other; p = 0.073, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

7. Secondary Outcome: Percentage of Patients With at Least One Episode of Significant Ketosis and/ or Risk Level for Impending Diabetic Ketoacidosis
Description: Diabetic ketoacidosis (DKA) is preceded by an increase in ketone production, resulting in blood ketone value increase (hyperketonemia) and later in ketone urine value (hyperketonuria).
  Significant hyperketonemia and risk level for impending diabetic ketoacidosis (DKA) are reported respectively as a blood ketone value from 0.6 to 1.5 mmol/L and >1.5 mmol/l
Time Frame: over 13 weeks of each treatment period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Insulin Glulisine | Insulin Aspart | Insulin Lispro
Number analyzed (Participants) | 256 | 256 | 256
percentage of patients | 17.6 [12.9 to 22.2] | 10.9 [7.1 to 14.8] | 11.7 [7.8 to 15.7]
Statistical Analysis 1: Comparison: Insulin Glulisine vs Insulin Aspart; Test type: Superiority or Other; p = 0.017, McNemar — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Insulin Glulisine vs Insulin Lispro; Test type: Superiority or Other; p = 0.032, McNemar — [p-value comment as in outcome 1, analysis 1]

8. Secondary Outcome: Monthly Rate of Episode of Significant Ketosis and/ or Risk Level for Impending Diabetic Ketoacidosis
Description: as for outcome 7
Time Frame: over 13 weeks of each treatment period
Population: as for outcome 1
Measure: Mean (Standard Error); unit: events per patient per month
Arm/Group | Insulin Glulisine | Insulin Aspart | Insulin Lispro
Number analyzed (Participants) | 256 | 256 | 256
events per patient per month | 0.14 (0.43) | 0.06 (0.22) | 0.06 (0.18)
Statistical Analysis 1: Comparison: Insulin Glulisine vs Insulin Aspart; Test type: Superiority or Other; p = 0.009, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Insulin Glulisine vs Insulin Lispro; Test type: Superiority or Other; p = 0.019, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

9. Secondary Outcome: Rate of Symptomatic Hypoglycemia With a Plasma Glucose (PG) ≤ 70 mg/dL Per Patient-year
Description: Symptomatic hypoglycemia is defined as an event with clinical symptoms that are considered to results from hypoglycemia (confirmed or not by a glucose measurement) and associated with prompt recovery after oral carbohydrate administration.
Time Frame: over 13 weeks of each treatment period
Population: as for outcome 1
Measure: Mean (Standard Error); unit: events in patient-year
Arm/Group | Insulin Glulisine | Insulin Aspart | Insulin Lispro
Number analyzed (Participants) | 256 | 256 | 256
events in patient-year | 73.88 (4.74) | 65.06 (4.74) | 62.74 (4.74)
Statistical Analysis 1: Comparison: Insulin Glulisine vs Insulin Aspart; Test type: Superiority or Other; p = 0.008, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Insulin Glulisine vs Insulin Lispro; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

10. Secondary Outcome: Rate of Severe Symptomatic Hypoglycemia Per Patient-year
Description: Severe symptomatic hypoglycemia is defined as an event with clinical symptoms that are considered to results from hypoglycemia in which the patient required assistance of another person and one of the following:
  * the event was associated with a measured blood glucose level below 36 mg/dL
  * or event was associated with prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration.
Time Frame: over 13 weeks of each treatment period
Population: as for outcome 1
Measure: Mean (Standard Error); unit: events in patient-year
Arm/Group | Insulin Glulisine | Insulin Aspart | Insulin Lispro
Number analyzed (Participants) | 256 | 256 | 256
events in patient-year | 1.63 (0.35) | 1.39 (0.35) | 1.07 (0.35)
Statistical Analysis 1: Comparison: Insulin Glulisine vs Insulin Aspart; Test type: Superiority or Other; p = 0.563, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Insulin Glulisine vs Insulin Lispro; Test type: Superiority or Other; p = 0.186, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

11. Secondary Outcome: Rate of Nocturnal Symptomatic Hypoglycemia With a Plasma Glucose (PG) ≤70 mg/dL Per Patient-year
Description: Nocturnal Symptomatic hypoglycemia was defined as an event with clinical symptoms that are considered to result from hypoglycemia (confirmed or not by a glucose measurement) and associated with prompt recovery after oral carbohydrate administration which occurs while the patient is asleep, after bedtime and before getting up in the morning.
Time Frame: over 13 weeks of each treatment period
Population: as for outcome 1
Measure: Mean (Standard Error); unit: events in patient-year
Arm/Group | Insulin Glulisine | Insulin Aspart | Insulin Lispro
Number analyzed (Participants) | 256 | 256 | 256
events in patient-year | 12.80 (0.95) | 9.66 (0.95) | 9.48 (0.95)
Statistical Analysis 1: Comparison: Insulin Glulisine vs Insulin Aspart; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Insulin Glulisine vs Insulin Lispro; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

12. Secondary Outcome: Patients With at Least One Site Infection, Site Inflammation/Erythema, Pruritus or Isolated Pain at Injection Site
Description: Infection: local reaction at the infusion site requiring local or systemic antibiotherapy, or local drainage as per Investigator judgment.
  Site inflammation or erythema: local reaction at the infusion site with no need for local or systemic antibiotherapy as per Investigator judgment.
  Pruritis at injection site: presence of pruritis at the infusion site without any symptom of inflammation or erythema and/or infection.
  Isolated pain at injection site: presence of pain at the infusion site without any symptom of inflammation or erythema and/or infection.
Time Frame: over 13 weeks of each treatment period
Population: as for outcome 1
Measure: Number; unit: patients
Arm/Group | Insulin Glulisine | Insulin Aspart | Insulin Lispro
Number analyzed (Participants) | 256 | 256 | 256
patients | 110 | 110 | 107
Statistical Analysis 1: Comparison: Insulin Glulisine vs Insulin Aspart; Test type: Superiority or Other; p = 1.000, McNemar — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Insulin Glulisine vs Insulin Lispro; Test type: Superiority or Other; p = 0.701, McNemar — [p-value comment as in outcome 1, analysis 1]

13. Secondary Outcome: Time Interval Between Infusion Set Changes: All Changes
Description: Patients treated with insulin pump have to change their infusion set regularly (i.e.change was recommended every 48h). The patients were asked to report any change of their infusion set and the reason for change (routine basis or because of occurrence of a specific event such as occlusion, unexplained hyperglycemia or adverse event).
  "All changes" include all the changes whatever the reason such as routine or requested by occurrence of events.
Time Frame: over 13 weeks of each treatment period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Insulin Glulisine | Insulin Aspart | Insulin Lispro
Number analyzed (Participants) | 254 | 254 | 254
hours | 69.1 (20.70) | 69.44 (19.22) | 69.98 (21.64)

14. Secondary Outcome: Time Interval Between Infusion Set Changes in Routine
Description: Patients treated with insulin pump have to change their infusion set regularly (i.e.change was recommended every 48h). The patients were asked to report any change of their infusion set and the reason for change (routine basis or because of occurrence of a specific event such as occlusion, unexplained hyperglycemia or adverse event).
  Changes in routine correspond to interval between changes according to patient use.
Time Frame: over 13 weeks of each treatment period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Insulin Glulisine | Insulin Aspart | Insulin Lispro
Number analyzed (Participants) | 254 | 254 | 254
hours | 70.72 (21.47) | 71.00 (20.68) | 71.07 (21.65)

15. Secondary Outcome: Glycosylated Hemoglobin: HbA1c
Description: Glycolysated Haemoglobin (HbA1c) is a biological parameter that reflects the blood glucose concentration over a long period of time. It is the standard parameter for glycemic control follow-up in diabetic patients. This parameter is expressed in percentage (%) and the target in diabetes management is to reach a HbA1c <7%
Time Frame: over 13 weeks of each treatment period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Insulin Glulisine | Insulin Aspart | Insulin Lispro
Number analyzed (Participants) | 256 | 256 | 256
percentage
  First week (week 1) (n=253, n=254, n=255) | 7.31 (0.71) | 7.33 (0.71) | 7.28 (0.71)
  Last week (week 13) (n=252, n=255, n=251) | 7.32 (0.03) | 7.25 (0.03) | 7.33 (0.03)
Statistical Analysis 1: Comparison: Insulin Glulisine vs Insulin Aspart; Test type: Superiority or Other; p = 0.078, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA adjusted on HbA1c value at the start of the first period
Statistical Analysis 2: Comparison: Insulin Glulisine vs Insulin Lispro; Test type: Superiority or Other; p = 0.938, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA adjusted on HbA1c level at the start of the first period

16. Secondary Outcome: Total Daily Basal Insulin Infusion
Description: dose of the basal insulin regimen administered throughout the 24-hour period
Time Frame: over 13 weeks of each treatment period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units
Arm/Group | Insulin Glulisine | Insulin Aspart | Insulin Lispro
Number analyzed (Participants) | 256 | 256 | 256
Units
  First week (week 1) (n=251, n=249, n=250) | 20.83 (9.05) | 20.93 (9.45) | 20.85 (9.16)
  Last week (week 13) (n=251, n=249, n=251) | 20.86 (9.24) | 20.81 (9.73) | 21.11 (9.38)

17. Secondary Outcome: Total Daily Bolus Insulin Dose
Description: dose of every increment administered for example before meals
Time Frame: over 13 weeks of each treatment period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units
Arm/Group | Insulin Glulisine | Insulin Aspart | Insulin Lispro
Number analyzed (Participants) | 256 | 256 | 256
Units
  First week (week 1) (n=249, n=247, n=250) | 18.63 (9.22) | 18.49 (9.00) | 18.40 (8.69)
  Last week (week 13) (n=248, n=244, n=249) | 18.58 (8.49) | 18.64 (9.60) | 19.19 (9.13)

ADVERSE EVENTS:
Time Frame: Adverse events are collected from the first to the last drug intake (3 periods x 13 weeks) + 1 week after the administration of the last intake i.e. end of the study.
Description: The safety analyses are performed on the safety population which includes all randomized and treated patients. Safety population is defined based on actual treatment received.
Arm/Group | Insulin Glulisine | Insulin Aspart | Insulin Lispro
Serious Adverse Events (participants affected / at risk) | 29/274 | 18/266 | 11/269
Other Adverse Events (participants affected / at risk) | 47/274 | 24/266 | 30/269
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Insulin Glulisine (N=274) | Insulin Aspart (N=266) | Insulin Lispro (N=269)
hypoglycaemic seizure (Metabolism and nutrition disorders) | 8 | 3 | 4
ketosis (Metabolism and nutrition disorders) | 9 | 4 | 2
hypoglycaemic unconsciousness (Metabolism and nutrition disorders) | 4 | 6 | 2
hypoglycaemia (Metabolism and nutrition disorders) | 3 | 0 | 0
diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
arteritis coronary (Cardiac disorders) | 0 | 1 | 0
cardiovascular disorders (Cardiac disorders) | 1 | 0 | 0
coronary artery stenosis (Cardiac disorders) | 0 | 1 | 0
myocardial infarction (Cardiac disorders) | 0 | 1 | 0
overdose (Injury, poisoning and procedural complications) | 1 | 1 | 0
forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
headache (Nervous system disorders) | 0 | 1 | 0
hemianopia (Nervous system disorders) | 0 | 0 | 1
hypoglycaemic coma (Nervous system disorders) | 0 | 1 | 0
chest pain (General disorders) | 1 | 1 | 0
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
depression (Psychiatric disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Insulin Glulisine (N=274) | Insulin Aspart (N=266) | Insulin Lispro (N=269)
Ketosis (Metabolism and nutrition disorders) | 47 | 24 | 30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.